CLINICAL TRIAL: NCT01496157
Title: Evaluation of PSMA-based PET as an Imaging Biomarker of Primary Prostate Cancer
Brief Title: Evaluation of Prostate-specific Membrane Antigen (PSMA)-Based PET Imaging of Primary Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: J1191; NA_00051395 (Other: JHMIRB)
Record Dates: First submitted 2011-12-13; First posted 2011-12-21 (Estimated); Results first posted 2018-08-28 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-07

CONDITIONS: Prostate Cancer
Keywords: Primary Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — N-(N-((S)-1,3-Dicarboxypropyl)carbamoyl)-4-(18F)fluorobenzyl-L-cysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patients with Primary Prostate Cancer (Experimental): Patients will be imaged with 18F-DCFBC
  Interventions: Drug: 18F-DCFBC

INTERVENTIONS:
Drug: 18F-DCFBC — A bolus of 10 mCi (370 MBq) [9-11 mCi (333-407 MBq)] of 18F-DCFBC will be injected into the IV line by slow IV push.

SUMMARY:
The objective of this study is to evaluate a radiolabeled urea-based small molecule inhibitor of prostate-specific membrane antigen (PSMA), [18F]DCFBC (DCFBC), as a PET imaging biomarker of prostate cancer detection and aggressiveness at initial diagnosis. PSMA is a well characterized histological marker of prostate cancer tumor aggressiveness but a quantitative non-invasive method for PSMA detection and monitoring is not currently available. Development of such an imaging biomarker would be useful to differentiate indolent from aggressive prostate cancer phenotypes and allow for selection of appropriate risk adaptive therapies. The investigators preliminary first-in-human studies demonstrate high specific DCFBC uptake in metastatic prostate cancer and feasibility for prostate cancer imaging. The investigators propose to study patients initially diagnosed with biopsy-positive prostate cancer to determine if DCFBC uptake and location by PET imaging will be positively correlated with prostate cancer by prostatectomy tissue step-section analysis. DCFBC uptake at sites of suspected metastatic disease will be compared to conventional imaging modalities (CT, bone scan) and biopsy results when available. In addition, DCFBC-PET uptake quantification will be compared with expression levels of PSMA and other prostate cancer relevant markers (PSA, Ki-67, TMPRSS2-ERG) by prostate tissue immunohistochemistry analysis and compared with clinical prognostic markers (PSA, Gleason score, clinical stage, Partin tables derived prediction of pathologic stage).

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed prostate cancer pathologically proven by prostate biopsy
2. Prostate biopsy histology grade ≥ Gleason 3+3=6.
3. Patients considered as candidates for and medically fit to undergo prostatectomy
4. At least 10 days after most recent prostate biopsy
5. No known problems with peripheral IV or central line access
6. Able to tolerate urinary straight catheter placement
7. Patient is judged by the Investigator to have the initiative and means to be compliant with the protocol and be within geographical proximity to make the required study visits.
8. Patients or their legal representatives must have the ability to read, understand and provide written informed consent for the initiation of any study related procedures.

Exclusion Criteria:

1. Prior pelvic external beam radiation therapy or brachytherapy
2. Chemotherapy for prostate cancer
3. Hormone deprivation therapy
4. Investigational therapy for prostate cancer
5. Hemorrhagic cystitis or active prostatitis
6. Unable to lie flat during or tolerate PET/CT
7. Prior history of any other malignancy within the last 2 years, other than skin basal cell or cutaneous superficial squamous cell carcinoma that has not metastasized and superficial bladder cancer
8. No prostatectomy scheduled prior to follow-up visit (12 to 72 hours post imaging)
9. Serum creatinine > 1.5 mg/dL or creatinine clearance < 50 mL/min/1.73m2

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-09-11 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2017-09-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven P Rowe, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Rowe SP, Gage KL, Faraj SF, Macura KJ, Cornish TC, Gonzalez-Roibon N, Guner G, Munari E, Partin AW, Pavlovich CP, Han M, Carter HB, Bivalacqua TJ, Blackford A, Holt D, Dannals RF, Netto GJ, Lodge MA, Mease RC, Pomper MG, Cho SY. (1)(8)F-DCFBC PET/CT for PSMA-Based Detection and Characterization of Primary Prostate Cancer. J Nucl Med. 2015 Jul;56(7):1003-1010. doi: 10.2967/jnumed.115.154336. Epub 2015 Jun 11. PMID 26069305

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2 enrolled participants were screen failures, therefore 13 started the study.
Period: Overall Study
Arm/Group | Patients With Primary Prostate Cancer
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients With Primary Prostate Cancer
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 13
Prostate specific antigen (PSA) [Mean (Standard Deviation); unit: ng/mL] | 8.36 (3.77)
Biopsy Gleason Score [Count of Participants; unit: Participants] — The Gleason score is an indication of prognosis based on prostate pathology. The total score ranges from 2 to 10 (ie: "1+1" to "5+5") with a higher score reflecting less-differentiated tumors with worse prognosis. The total score is a sum of two numbers which are based on the microscopic appearance of cells. The first number is the score based on the dominant, cell morphology (scored 1-5) and the second number is based on the highest grade of the non-dominant cell pattern (scored 1-5).
  Participants
    Gleason score 3+3 | 1
    Gleason Score 3+4 | 5
    Gleason Score 4+3 | 4
    Gleason Score 4+4 | 3
Prostatectomy gleason score [Count of Participants; unit: Participants] — The Gleason score is an indication of prognosis based on prostate pathology. The total score ranges from 2 to 10 (ie: "1+1" to "5+5") with a higher score reflecting less-differentiated tumors with worse prognosis. The total score is a sum of two numbers which are based on the microscopic appearance of cells. The first number is the score based on the dominant, cell morphology (scored 1-5) and the second number is based on the highest grade of the non-dominant cell pattern (scored 1-5).
  Participants
    Gleason 3+3 | 1
    Gleason 3+4 | 5
    Gleason 4+3 | 2
    Gleason 4+4 | 1
    Gleason 4+5 | 3
    Gleason 5+3 | 1

OUTCOME MEASURES:

1. Primary Outcome: PET Detection of Primary Prostate Cancer
Description: To compare number of participants with positive or negative uptake of 18F-DCFBC in primary prostate cancer by DCFBC PET to prostatectomy pathology as determined by tissue step-section analysis in men with biopsy-positive prostate cancer (Gleason score > 4+3=7).
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Primary Prostate Cancer
Number analyzed (Participants) | 13
Participants
  Prostate Cancer with Positive Uptake of 18F-DCFBC | 6
  Prostate Cancer with Negative Uptake of 18F-DCFBC | 7

2. Secondary Outcome: PET Detection of Metastatic Disease at Initial Staging
Description: To compare the detection of bone and nodal metastatic disease by DCFBC PET at initial staging to detection by available conventional imaging modalities (bone scan, CT, MRI) and biopsy pathology.
Time Frame: 24 months
Population: Data was not collected for this outcome measure.
Arm/Group | Patients With Primary Prostate Cancer
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 3 years
Arm/Group | Patients With Primary Prostate Cancer
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No